CLINICAL TRIAL: NCT01038258
Title: Monitoring Response After The First Chemotherapy Cycle In Newly Diagnosed Breast Cancer As A Guide For Neoadjuvant Therapy
Brief Title: Monitoring Response After The First Chemotherapy Cycle After Neoadjuvant Breast Cancer Therapy
Acronym: PETBreast
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Auxilio Mutuo Cancer Center (Other)
Collaborators: Sononuclear (Unknown)
Responsible Party: Principal Investigator, Fernando Cabanillas, Hematology-Oncologist, Auxilio Mutuo Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCAM 07
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Invasive Ductal Carcinoma; Lobular Breast Carcinoma; Inflammatory Breast Carcinoma
Keywords: neoadjuvant chemotherapy
MeSH Terms: conditions — Carcinoma, Lobular; Inflammatory Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- No arms (Other): No arms
  Interventions: Procedure: PET scan after course 1 and surgery after 8 courses

INTERVENTIONS:
Procedure: PET scan after course 1 and surgery after 8 courses — PET scan and surgery

SUMMARY:
A PET scan drop less than 20% in SUVs or below a certain absolute SUV value after the first course of neoadjuvant chemotherapy can predict pathological response, and could in the future lead to an early surgical intervention.

DETAILED DESCRIPTION:
The use of neo-adjuvant systemic therapy in women recently diagnosed with breast cancer is growing in popularity based on its proven benefit (1). Pre-operative chemotherapy not only can assist in regards to breast conservation therapy (2) but data suggest prognostic benefits in those subset of patient's obtaining complete pathological response (3,4) .

It is imperative for clinicians to detect as early as possible those patients likely to obtain the desired clinical and /or pathologic response, thus identifying those patients who don't benefit from the first line neoadjuvant treatment so that their treatment can be modified accordingly.

Response to treatment based on clinical data or structural imaging, usually requires several chemotherapeutic cycles to establish degree of effectiveness (5). Lately, FDG-PET/CT has been used in different types of neoplasms, breast cancer among them, to establish early response to treatment (6,7). Recent data has established the usefulness of metabolic analysis via FDG-PET, in separating subgroups of chemotherapy. For such analytical approach, sequential estimation of SUVs (Standardized Uptake Value) have been measured along the duration of the treatment. Reduction in SUVs presumes adequate response to treatment (8), while little or no change in metabolic activity presumes sub-optimal response .

However, no definite consensus has been established in regards to what degree of metabolic response is predictive of the desired clinical benefit, particularly early in the treatment . Establishing such criteria could potentially serve as a guideline for monitoring neoadjuvant treatment. Schelling et al, was able to separate a group of patients that eventually showed either progression of the disease or no clinical response as early as the first course of chemotherapy.

The aim of our study is to establish a simple formula using FDG-PET/CT, as early as the first course of chemotherapy, to stratify patients undergoing neoadjuvant chemotherapy for recently diagnosed breast cancer. Those who will benefit from continuing the same treatment will be regarded as responders versus non-responders, which are those in need of changing strategy.

The primary goal of this study is to correlate the results of FDG-PET/CT performed 15 days after the first course of chemotherapy versus those of clinical assessment and breast MRI obtained after the 3rd course of chemotherapy. At that time, a clinical decision on which therapeutic path to be followed will be made.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed breast carcinoma that will receive neoadjuvant chemotherapy based on: Tumors size greater than 2 cms; Locally advanced tumors, Tumors close to or invading chest wall or areola and/or Inflammatory Breast cancer.
* 18 years of age.
* Available for follow-up visits
* Able to comply with study requirements.
* Have signed an IRB approved written informed consent form

Exclusion Criteria:

* Any significant medical or psychiatric illness, which would prevent the patient from giving informed consent or following the study procedures.
* Pregnant and Nursing women.
* No restriction will be placed on the chemotherapy regimen used although we expect that most patients will receive Anthracycline based regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-07; Primary Completion 2011-12 (Actual); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Pathologic response | After 1st course of chemo and after definitive surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Cabanillas, MD, Principal Investigator — Hospital Auxilio Mutuo Cancer Center
Locations (1):
- Hospital Auxilio Mutuo Cancer Center, San Juan, Puerto Rico, Puerto Rico